CLINICAL TRIAL: NCT00002410
Title: A Phase III, Multicenter, Randomized, Open-Label Study to Compare Antiretroviral Activity and Tolerability of Three Different Combination Regimens (DMP 266 + Indinavir, DMP 266 + Zidovudine + Lamivudine, Indinavir + Zidovudine + Lamivudine) in HIV-Infected Patients
Brief Title: A Study of Three Different Anti-HIV Drug Combinations in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dupont Merck (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 281B; DMP 266-006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Drug Resistance, Microbial; HIV Protease Inhibitors; Lamivudine; Indinavir; Genotype; Reverse Transcriptase Inhibitors; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of three anti-HIV drug combinations. The three combinations are: (1) efavirenz (DMP 266) plus indinavir; (2) DMP 266 plus zidovudine (ZDV) plus lamivudine (3TC); and (3) indinavir plus ZDV plus 3TC. This study also examines the resistance HIV may have to these drugs and if these drugs are effective over a long period of time.

ELIGIBILITY:
Exclusion Criteria

Concurrent Medication:

Excluded:

* Terfenadine, astemizole, cisapride, triazolam, or midazolam (competition for the enzyme cytochrome P-450 3A4 [CYP3A4] by indinavir could result in inhibition of metabolic breakdown of these drugs and create the potential for serious and/or life threatening events [i.e., cardiac arrhythmia, prolonged sedation]).
* Rifampin or rifabutin (prohibited because of potential drug interaction with indinavir).
* Ketoconazole, itraconazole, and clarithromycin.
* Concomitant systemic therapy for acute opportunistic infection or malignancy.

Excluded:

Life expectancy less than 12 months.

Prior Medication:

Excluded:

* Prior treatment with efavirenz, 3TC, an NNRTI, or an HIV protease inhibitor.
* Prior antiretroviral agent within 14 days of initiating study treatment.
* Prior treatment (within 30 days of initiating study treatment) with any other experimental drug for any indication.

Patients must:

* Have a diagnosis of HIV infection.
* Have CD4 counts greater than or equal to 50 cell/mm3.
* Have a life expectancy greater than or equal to 12 months.
* Be post-pubescent.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (41):
- United States (40):
  - Phoenix Body Positive, Phoenix, Arizona
  - Arizona Clinical Research Ctr Inc, Tucson, Arizona
  - Richard Stryker, Beverly Hills, California
  - Paul Cimoch, Irvine, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Kraus Med Group, Los Angeles, California
  - Oasis Clinic / Martin Luther Jr Gen Hosp / King-Drew Med Ctr, Los Angeles, California
  - Blick Med Associates, Stamford, Connecticut
  - Novum Inc, Washington D.C., District of Columbia
  - Bach and Godofsky, Bradenton, Florida
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Boulevard Comprehensive Care Ctr, Jacksonville, Florida
  - Larry Marc Bush / c/o Sally Yantis, Lake Worth, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Ctr for Quality Care, Tampa, Florida
  - Daniel Seekins, Tampa, Florida
  - Infectious Disease Research Institute, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Georgia Research Associates, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Infectious Diseases, Indianapolis, Indiana
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Univ of Nebraska Med Ctr / HIV Clinic, Omaha, Nebraska
  - Univ Med Ctr / HIV Wellness Ctr, Las Vegas, Nevada
  - Community Research Initiative on AIDS, New York, New York
  - Clinical Directors Network / HIV/AIDS Program Manager, New York, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Remington-Davis Inc, Columbus, Ohio
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - The Miriam Hosp, Providence, Rhode Island
  - Research Services 2000 Inc, Dallas, Texas
  - Division of Infectious Disease / Dept of Internal Medicine, Dallas, Texas
  - Research Services 2000 Inc, Fort Worth, Texas
  - Montrose Clinic, Houston, Texas
  - UT-Health Science Ctr, Houston, Texas
  - Diagnostic Clinic of San Antonio, San Antonio, Texas
  - Oyster Point Med Specialists, Newport News, Virginia
  - Novum Inc / Pharmaceutical Research Services, Seattle, Washington
  - Infectious Diseases Associates, Milwaukee, Wisconsin
- Javier O Morales Ramirez, San Juan, Puerto Rico